CLINICAL TRIAL: NCT04331483
Title: A Feasibility Study to Assess Connected Bikes as a Means of Adapted Physical Activity in Children, Adolescents and Young Adults Requiring Hematopoietic Stem Cell Allografts
Brief Title: A Study to Assess a Physical Activity Program in Children, Adolescents and Young Adults Requiring Hematopoietic Stem Cell Allografts
Acronym: EVAADE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: modification of the intervention before patient's enrollment, new protocol submitted
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EVAADE; ET 18-184 (Other: Sponsor ID)
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Haematological Malignancy; Acute Leukemia; Myelodysplastic Syndromes; Hemoglobinopathy in Children; Bone Marrow Aplasia; Severe Combined Immunodeficiency
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Anemia, Aplastic; Severe Combined Immunodeficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity intervention (Experimental): The intervention consists of an adapted physical activity (APA) program defined at baseline, incorporating supervised sessions with an APA teacher, as well as autonomous sessions. The program is individualized according to age, aerobic capacity, and PA preferences.
  The total duration of the intervention is a maximum of 3 months (during the period of hospitalization in a sterile room).
  Interventions: Other: Physical activity program

INTERVENTIONS:
Other: Physical activity program — Supervised sessions of at least 15 minutes 4 times a Week combined with unsupervised sessions.
  The supervised activities include moderate-intensity aerobic activities (exercise bike), muscle strengthening (dumbbells, elastic bands, medicine balls) and playful situations (ball games, cooperative games, body expression games).
  Each patient can also do unsupervised sessions, autonomously, on the bike thanks to a smartphone application developed by the Kiplin company, with challenges to be carried out by teams of 2 to 5 people (team including several patients, possibility to include relatives) over periods of 1 to 3 weeks per challenge.

SUMMARY:
To date, allogeneic haematopoietic stem cell transplantation (aHSCT) is the only curative treatment for many paediatric and young adult haematological pathologies (acute leukaemia, myelodysplastic syndromes, haemoglobinopathies, bone marrow aplasia, severe combined immunodeficiency). Despite the major therapeutic progress made over the last 50 years, particularly in terms of supportive care, post-transplant morbidity and mortality remains high. Infectious complications, whose incidence varies between 30 and 60%, are the first cause of mortality in the immediate post-transplant period.

In order to protect the patient from the occurrence of severe infectious episodes, aHSCTmust be performed in a highly protected environment (positive pressure chambers).

This has implications for the experience and impact of hospitalization on the patient and family. This is particularly true in paediatrics, whether in children, adolescents or young adults, where it is not only the patient's quality of life that is at stake, but also their emotional and psychomotor development. In these patients, prolonged hospitalization (at least 6 weeks) in a sterile room will be responsible for physical deconditioning accompanied by a decrease in muscle mass, itself concomitant with undernutrition, and an increase in sedentary lifestyle. This prolonged hospitalisation in a sterile room, associated with myeloablative treatments, is therefore the cause of social isolation of patients, but it is also often synonymous with physical inactivity leading to a rapid decrease in physical condition, quality of life and an increase in fatigue.

Today, the benefits of physical activity (PA) during and after cancer treatment have been widely demonstrated.

The objective is to evaluate the feasibility of an adapted physical activity program during the isolation phase for achieving aHSCT in children, adolescents and young adults. This is a prospective, interventional, monocentric cohort study conducted at the Institute of Paediatric Haematology and Oncology in Lyon. The intervention will take place during the isolation phase and consists of an adapted physical activity (APA) program defined at inclusion, integrating supervised sessions with an APA teacher, as well as autonomous sessions. The program is individualized according to age, aerobic capacity, and PA preferences. Sessions are also tailored to the biological, psychological, and social parameters of patients.

The total duration of the intervention is 3 months. To date, no PA studies have been performed in patients under 21 years of age requiring aGCSH during the sterile isolation phase. EVAADE will therefore be the first study in this population to offer an innovative procedure with a connected device.

ELIGIBILITY:
Inclusion Criteria:

* 8 years ≤ Age ≤ 21 years
* Size more or equal to 110 cm.
* Histologically or cytologically confirmed malignant or non-malignant haemopathy
* Indication for hematopoietic stem cell allograft.
* Hospitalization in a protected room at IHOP/DAJAC.
* Certificate of no contraindication to the practice of an APA, issued by the oncologist or attending physician.
* Having available in the sterile room a smartphone (iPhone 5S version for Apple/version 5 under Android at least) or a tablet (for the realization of the connected challenges) during the whole hospitalization period.
* Written consent signed and dated by the patient or the parents of minor patients with the acceptance of the minor.

Exclusion Criteria:

* Severe Heart Disease and Uncontrolled Cardiovascular Disease

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-08 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Observance to the physical activity program | weekly from baseline to 3 months
  achieved/non-achieved (achived meaning the patient attended at least one session of 15 minutes weekly during the whole program

SECONDARY OUTCOMES:
Impact of the physical activity program on weight | Baseline, 1 month and 3 months
  weight in kgs
Impact of the physical activity program on waist circumference | Baseline, 1 month and 3 months
  assessed in cm
Impact of the physical activity program on hip circumference | Baseline, 1 month and 3 months
  assessed in cm
Impact of the physical activity program on abdominal circumference | Baseline, 1 month and 3 months
  assessed in cm
Impact of the physical activity program on body mass index | Baseline, 1 month and 3 months
  weight/(size)2
Impact of the physical activity program on endurance capacity | Baseline, 1 month and 3 months
  Harvard step test
Impact of the physical activity program on muscle strength | Baseline, 1 month and 3 months
  Dynamometer
Impact of the physical activity program on fatigue | Baseline, 1 month and 3 months
  Visual analogic scale from 0 to 10
Self-efficacy feeling | 3 months
  HAPA questionnaire
Motivation towards physical activity | Baseline, 1 month and 3 months
  BREQ questionnaire
Impact of the PA program on metabolic syndrome | Baseline and 3 months
  Lipid check-up

CONTACTS AND LOCATIONS:
Overall Officials: Carine HALFON-DOMENECH, MD, Principal Investigator — Institut d'Hematologie et d'Oncologie Pédiatrique
Locations (1):
- Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon, France

IPD SHARING:
Plan to Share IPD: No